CLINICAL TRIAL: NCT00824317
Title: Stimulant Drug Treatment of AD/HD, Inattentive Type
Brief Title: Stimulant Drug Treatment of Attention-Deficit Hyperactivity Disorder (AD/HD), Inattentive Type
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Mary Solanto, Associate Professor, Mount Sinai School of Medicine
Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-0394; R21MH062945 (NIH)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): methylphenidate
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: methylphenidate — (15 mg daily), medium (25 mg daily) and high (40 mg daily)
  Arms: 2
Drug: Placebo
  Arms: 1

SUMMARY:
The purpose of this study is to compare the response to methylphenidate treatment of children with two different subtypes of ADHD.

DETAILED DESCRIPTION:
The Inattentive subtype (IN) of Attention-Deficit/Hyperactivity Disorder was newly defined in DSM-IV (1994). Recent epidemiological studies suggest that IN is at least as common and as impairing academically and socially as the more commonly recognized Combined type (CB). However, little is known about the etiology, course and outcome, or treatment of the IN type. Notably, although stimulant drugs are commonly used clinically to treat the disorder, there have been no systematic studies of its efficacy in the IN subtype. Differences between the IN and CB subtypes in behavioral phenotype, as well as in gender ratio, age of onset, and comorbidity suggest there may be critical differences in neurobiology, which may have relevance for response to drug treatments. The lack of data concerning stimulant drug efficacy in the IN type thus constitutes an important issue from the perspective of public health and quality of care. The proposed research is responsive to the current RFA in that it will study the efficacy of an established treatment (stimulants) in a new patient population (the IN subtype). A second specific aim is to test a hypothesis, emerging from a review of the literature, of divergence between dose-response curves for effects on activity and attention. We predict that the dose that optimizes performance on ratings of hyperactivity-impulsivity will be lower than that which optimizes performance on ratings of academic function and on the neuropsychological tests. We will similarly examine whether differences in dose-response curves for specific functions extend to differences between subtypes in optimal dose. The final aim of the current study is to compare the IN and CB subtypes with respect to selected measures of neurocognitive function on placebo and in response to drug treatment. We predict that the IN subtype will perform more poorly on measures of spatial orienting and stimulus encoding, whereas the CB subtype will show greater deficits on measures of cognitive inhibitory control, and that both types of cognitive deficit will respond to drug treatment.

ELIGIBILITY:
Inclusion Criteria:Inattentive Subtype:

Inclusion Criteria:

1. A diagnosis on the structured DISC interview conducted with the parent, of ADHD, Predominantly Inattentive Type.
2. Ratings by parent and by teacher corresponding to a total score above the 93rd percentile (i.e. more than 1.5 SD above the mean) on the scale of "DSM-IV Inattention" on the current Conners Parent (or Teacher) Rating Scale - Long Form. The items on this scale are the inattention symptom criteria from the DSM-IV, each of which the informant is asked to rate in severity on a 4-point scale ranging in severity from 0 ("not at all") to 3 ("very much"). A score above the 93th percentile indicates that the child's score equals or exceeds that for 93% of other children of the same age (within 2 years) and gender.

Exclusion Criteria:

(a) Scores more than 1 SD (84th percentile) above the mean on the DSM-IV-Hyperactive-Impulsive scale on the Conners Parent or Teacher Rating Scales-Long Form.

Combined Subtype:

Inclusion Criteria:

1. A diagnosis of ADHD, Combined type on the structured DISC interview with the parent.
2. Ratings by parent and teacher each corresponding to a total score above the 93rd percentile (i.e. more than 1.5 SD above the mean) on the scale of "DSM-IV attention" on the current Conners Parent (Teacher) Rating Scales - Long Form.
3. Ratings by parent and teacher each corresponding to a total score above the 93rd percentile (i.e. more than 1.5 SD above the mean) on the scale of "DSM-IV Hyperactive-Impulsive" symptoms on the current Conners Parent (Teacher) Rating Scales - Long Form.

Both Groups:

Inclusion Criterion: The child's school must agree to administer medication at mid-day and to allow the teacher to complete the requisite behavior ratings.

Exclusion Criteria:

1. WISC-III full-scale IQ less than 80.
2. Major acute or chronic medical condition, including sensory loss, and neurological disorder, or any medical condition that would preclude the use of stimulant medication.
3. Comorbidity: The study rationale for inclusion/exclusion of comorbid psychological/psychiatric conditions is as follows: children for whom the study treatment is contraindicated, or for whom treatment not provided in the study is required immediately, will not be entered in the trial. Thus, as an example, comorbid depression or anxiety disorder is permitted provided immediate treatment of the depressive or anxiety disorder is not required. Tic disorders of mild to moderate severity, and stable, would be eligible for inclusion, as this would not constitute a contraindication to receiving stimulants. However, children with pronounced or unstable tics would not be eligible for the trial.

   Children with any of the following conditions will be excluded from the study: psychosis, any pervasive developmental disorder, and bipolar disorder. Thus children will be permitted in the study if they have a comorbid learning disability, oppositional defiant disorder, or conduct disorder. The Wechsler Individual Achievement Tests will be administered in order that we can characterize our sample with respect to the presence of comorbid learning disabilities.
4. Concomitant medications: Systemically absorbed medication will be exclusionary, while non-systemically absorbed medications will generally be permitted. Children who have taken any experimental medication in the past month will be excluded. Any prior psychotropic medication must have a suitable washout period of at least 4 half-lives before assessment can begin (generally a minimum of 2 weeks; up to 4 weeks for fluoxetine). Children taking methylphenidate at the time of inquiry may be withdrawn from medication only if treatment response is less than optimal and a re-evaluation is deemed clinically necessary. Children taking other psychotropic medication may be discontinued, provided their prescribing physician is in agreement with this plan, and provided there is clinical indication for doing so (i.e., either inadequate response, adverse effects or problematic time-action properties).

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2001-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
(BLIND) CLINICIAN RATING ON ADHD-RS (SYMPTOM CHECKLIST) AND CGI (CLINICAL GLOBAL IMPRESSIONS) | Weekly

SECONDARY OUTCOMES:
WEEKLY RATINGS BY PARENTS AND TEACHERS ON WELL-NORMED MEASURES OF ADHD SYMPTOMS AND FUNCTIONAL IMPAIRMENT PREVIOUSLY SHOWN TO BE DRUG-SENSITIVE (CONNERS AND SKAMP SCALES). | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Mary Solanto, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States